CLINICAL TRIAL: NCT04058756
Title: An Open-label, Multi-center Rollover Protocol for Continued Characterization of Safety and Tolerability for Subjects Who Have Participated in a Novartis-sponsored Spartalizumab Study as Single Agent or in Combination With Other Study Treatments
Brief Title: Rollover Study for Continued Safety and Tolerability in Subjects Treated With Spartalizumab Alone or in Combination With Other Study Treatments
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001X2X01B
Record Dates: First submitted 2019-08-13; First posted 2019-08-16 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors
Keywords: Phase Ib; PDR001; PD-1; continued access
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PDR001 (Experimental): All subjects in all combination will be entered in one arm
  Interventions: Drug: PDR001

INTERVENTIONS:
Drug: PDR001 — PDR001

SUMMARY:
The purpose of this study is to continue to assess safety and tolerability, and to allow continued access to study treatment for subjects already receiving spartalizumab as single agent or in combination with other study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subject is currently enrolled in a pre-defined Novartis-sponsored study and is receiving spartalizumab as single agent or in combination with other study treatment,
* Subject is currently deriving clinical benefit from the study treatment, as determined by the investigator.

Other protocol defined inclusion criteria may apply

Exclusion Criteria:

* Subject has been permanently discontinued from spartalizumab in the parent protocol for any reason other than enrollment in the Roll over Study
* Subject does not meet the criteria specified in the parent protocol criteria for continued study treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and nature of AE and SAE by subject | 5 years
  Safety data.
Number of subjects with PDR001 dose interruption and/or reduction | 5 years

SECONDARY OUTCOMES:
Number of subjects receiving PDR001 | 5 years
Subject's exposure duration | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- United States (3):
  - Columbia University Medical Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - MD Anderson Cancer Center Uni of Te, Houston, Texas
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- China (2):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Guangzhou
- Novartis Investigative Site, Brno, Czechia
- France (4):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Villejuif
- Germany (4):
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Ulm
- Hong Kong (3):
  - Novartis Investigative Site, High West
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Pokfulam
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Italy (6):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Leiden, South Holland, Netherlands
- Poland (2):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Poznan
- Novartis Investigative Site, Seoul, South Korea
- Spain (5):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Zurich, Switzerland
- Novartis Investigative Site, Taipei, Taiwan
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai